CLINICAL TRIAL: NCT04562090
Title: A Phase 4, Open-label, Randomized, Prospective, Interventional Post-authorization Efficacy and Safety Study of Mirabegron 50 mg and 25 mg for the Treatment of Overactive Bladder in Chinese Subjects
Brief Title: A Study With Mirabegron 50 mg and 25 mg in Chinese Participants With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 178-MA-2295; CTR20202160 (Registry Identifier: chinadrugtrials.org.cn)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Urge Incontinence; Overactive Bladder (OAB)
Keywords: mirabegron
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Participants fulfilling the screening inclusion/exclusion criteria were randomized in a 2:1 ratio, 50 mg mirabegron and 25 mg mirabegron, using a computer-generated randomization to reduce selection bias.
Masking Description: This was an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mirabegron 25 mg (Experimental): Participants received single oral dose of Mirabegron 25 milligrams (mg) tablet once daily, at the same time after a meal for a duration of 12 weeks. Dose escalation to 50 mg was permitted at Visit 3 (Week 4) or Visit 4 (Week 8) at the discretion of investigator.
  Interventions: Drug: mirabegron
- Mirabegron 50 mg (Experimental): Participants received single oral dose of Mirabegron 50 mg tablet once daily, at the same time after a meal for a duration of 12 weeks.
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — Mirabegron was administered as single oral dose of 25 mg or 50 mg sustained-release tablet
  Other Names: Betmiga

SUMMARY:
The purpose of this study was to evaluate the efficacy of mirabegron for the treatment of overactive bladder (OAB) in Chinese participants. This study also evaluated the safety of mirabegron for the treatment of OAB in Chinese participants, evaluated other efficacy variables of mirabegron for the treatment of OAB and explored different mirabegron starting doses.

DETAILED DESCRIPTION:
The study followed an open-label, randomized, 12-week, prospective, interventional post-authorization design for the treatment of OAB in 249 Chinese participants. Each eligible participant took part in a 12-week treatment period. Treatments were administered once daily orally after a meal during a 12-week, open-label treatment period. Study visits took place at weeks 4, 8 and 12. For the 25 mg mirabegron group, a dose escalation to 50 mg was permitted on visit 3 and visit 4 at the investigators' discretion. 15 study sites across China enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant should exhibit symptoms of OAB for at least 12 weeks before initiation of the screening period.
* Participant should have an average of ≥ 8 micturitions/24 hours.
* Participant should have an average of ≥ 1 episode of grade 3 or 4 (PPIUS) urgency or urgency incontinence/24 hours, during a 3-day micturition diary period.
* Female participant is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final investigational product (IP) administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
* Female participant must not donate ova starting at first dose of investigational product (IP) and throughout the study period and for 30 days after final IP administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and 30 days after final IP administration.
* Male participant must not donate sperm during the treatment period and for 30 days after final IP administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final IP administration.
* Participant agrees not to participate in another interventional study while participating in the present study, defined as 28 days prior screening until completion of the last study visit.

Exclusion Criteria:

Exclusion at Visit 1/Week -2 (Screening)

* Participant has stress urinary incontinence as a predominant symptom.
* Participant has an average total daily urine volume > 3000 mL (as recorded in a 3-day voiding diary period).
* Participant has indwelling catheter or practices intermittent self-catheterization.
* Participant has neurogenic detrusor overactivity or indicated pathology other than OAB.
* Participant as monosymptomatic enuresis.
* Participant has post void residual (PVR) volume of ≥ 100 mL or a clinically significant lower urinary tract obstructive disease, except if successfully treated.
* Participant has anatomical anomalies (surgically treated or untreated) that affect lower urinary tract function.
* Participant with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
* Participant has lower urinary tract stones or clinically significant kidney stones requiring treatment.
* Participant has interstitial cystitis.
* Participant has suffered from chronic urinary tract infection (UTI) or has had more than 3 ETIs in the 2 months prior to visit 1/week -1 to -2 (screening).
* Participant has uncontrolled hypertension (sitting systolic blood pressure [SBP] ≥ 180 mmHg or diastolic blood pressure [DBP] ≥ 110 mmHg).
* Participant has pulse rate ≥ 110 beats per minute (bpm) or <50 bpm.
* Participant has corrected QT interval by Fredericia (QTcF) > 440 msec on screening ECG or a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS] or family history of LQTS or exercise-induced syncope).
* Participant's aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is ≥ 2 × upper limit of normal (ULN) or total bilirubin (TBL) is ≥ 1.5 × ULN according to age and sex (participants with Gilbert's syndrome are excepted from the bilirubin threshold).
* Participant has moderate or severe renal impairment.
* Participant has a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) UTI. Note: if the UTI is treated successfully (clinical recovery: confirmed by dipstick test and repeated dipstick test after 14 days [both should be negative]), the participant can be rescreened.
* Participant has a history or presence of any malignancy (previous or current diagnosis of bladder or prostate cancer).
* Participant uses any drugs that are sensitive cytochrome P450 2D6 (CYP2D6) substrates with a narrow therapeutic index or sensitive P-glycoprotein (P-gp) substrates after the start of washout.
* Participant is using or has used prohibited prior and/or concomitant medication(s). In case α1-AR antagonists, 5α-reductase inhibitors (5-ARIs) and Phosphodiesterase type 5 inhibitors (PED-Is) are used for Benign Prostatic Hyperplasia(BPH), participant can be included in the study.
* Participant has known or suspected hypersensitivity to mirabegron or any components of the formulations used.
* Participants previously treated for OAB including medication and nondrug treatment. If the treatment stopped for 2 weeks or more prior to the screening visit, participants can be included in the study.
* Participant has participated in another clinical study (and/or participant has received any investigational therapy within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/week -1 to -2 (screening).
* Participant has constipation as defined by the Rome IV criteria that cannot be successfully treated prior to study entry.
* Female participant who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
* Participants has a positive serology test for hepatitis A virus (HAV) antibodies (immunoglobulin M [IgM]), hepatitis B core (HBc) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, antibodies to human immunodeficiency virus (HIV) or syphilis at screening.
* Participant is an employee of Astellas, the study-related contract research organizations (CROs) or the clinical unit.
* Participant has any condition which makes the participant unsuitable for study participation.

Additional Exclusion at Visit 2/Week 0 (Baseline)

* Participant has stress urinary incontinence as a predominant symptom.
* Participant has an average total daily urine volume > 3000 mL (as recorded in a 3-day voiding diary period).
* Participant has monosymptomatic enuresis confirmed by the bladder e-diary.
* Participant suffers from a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) UTI. Note: if a symptomatic UTI is present, all visit 2/week 0 (baseline) assessments must be postponed until the UTI is successfully treated (clinical recovery: confirmed by dipstick test and repeated dipstick test after 14 days [both should be negative]). The postponed visit 2/week 0 (baseline) should be within 14 days of the intended visit 2/week 0 (baseline).
* Participant with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
* Participant has uncontrolled hypertension (sitting SBP ≥ 180 mmHg or DBP ≥ 110 mmHg).
* Any reason that makes the participant unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Director, Study Director — Astellas Pharma China, Inc.
Locations (15):
- China (15):
  - Site CN86020, Wuhan, Hubei
  - Site CN86001, Beijing
  - Site CN86004, Beijing
  - Site CN86014, Beijing
  - Site CN86010, Chengdu
  - Site CN86009, Guangzhou
  - Site CN86018, Guangzhou
  - Site CN86003, Lanzhou
  - Site CN86013, Shanghai
  - Site CN86002, Suzhou
  - Site CN86021, Taiyuan
  - Site CN86011, Wuhan
  - Site CN86022, Wuxi
  - Site CN86012, Xi'an
  - Site CN86007, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=15079&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/178-MA-2295/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in China.
Pre-assignment Details: Participants with symptoms of overactive bladder (OAB) for at least 12 weeks before initiation of the screening period and who met all of the inclusion and none of the exclusion criteria were enrolled in this study.
Period: Overall Study
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Started | 84 | 165
Participants (Never-Up Titrated) | 44 | 0
Participants (Up Titrated to 50 mg) | 39 | 0
Treated | 83 | 165
Completed | 78 | 153
Not Completed | 6 | 12
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 2 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 1 | 4
Not completed — Miscellaneous | 0 | 3

BASELINE CHARACTERISTICS:
Population: All Randomized Set consisted of all participants who were randomized and had a randomization number.
Groups:
- Mirabegron 25 mg: Participants received single oral dose of mirabegron 25 mg tablet once daily, at the same time after a meal for a duration of 12 weeks. Dose escalation to 50 mg was permitted at Visit 3 (Week 4) or Visit 4 (Week 8) at the discretion of investigator.
- Total: Total of all reporting groups
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg | Total
Number analyzed (Participants) | 84 | 165 | 249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (16) | 50.6 (14.6) | 49.7 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 120 | 185
  Male | 19 | 45 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 84 | 165 | 249
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese Ethnicity | 84 | 165 | 249
Mean Number of Micturitions per 24 hours [Mean (Standard Deviation); unit: micturitions per 24 hours] — Population: Full Analysis Set included all participants who were randomized and received at least 1 dose of investigational product (IP) and had at least 1 post baseline measurement for mean number of micturitions per 24 hours. Participants with available data were analyzed.
  micturitions per 24 hours
    number analyzed (Participants) | 79 | 165 | 244
    (all) | 11.8 (6.36) | 11.77 (5.47) | 11.78 (5.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) to the End of 12-Week Treatment Period in Mean Number of Micturition/24 Hours in Mirabegron 50 mg Group
Description: A micturition was defined as any voluntary act of passing urine (excluding incontinence only episodes). The mean number of micturitions per 24 hours was calculated as the average number of times a participant urinated per day during the 3-day micturition diary period.
Time Frame: Baseline, week 12
Population: Full Analysis set (FAS) included all participants who were randomized and received at least 1 dose of investigational product (IP) and had at least 1 post baseline measurement for mean number of micturitions per 24 hours. Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Mirabegron 50 mg
Number analyzed (Participants) | 147
micturitions per 24 hours | -3.76 (0.40)
Statistical Analysis 1: Comparison: Mirabegron 50 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — Repeated Measures Analysis (RMA): CFB as response, treatment group (TG), visit (week 4, 8 and 12), pooled site, sex and the interaction between TG and visit as fixed effects and mean number of micturitions per 24 hours at baseline as covariate; LS Mean = -3.73, 95% CI 2-sided [-4.30 to -3.16], Standard Error of Mean 0.29

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: AE was defined as any untoward medical occurrence in a participant administered a study drug or had undergone study procedures and which did not necessarily have had a causal relationship with the treatment. An abnormality identified during a medical test (e.g., laboratory parameter, vital sign, Electrocardiography (ECG) data, and physical exam) was defined as an AE only if the abnormality induced clinical signs or symptoms or requires active intervention or requires interruption or discontinuation of study medication or the abnormality or investigational value was clinically significant in the opinion of the investigator. Treatment emergent AE was defined as an AE observed after starting administration of the IP and 30 days after the final administration of study drug.
Time Frame: From first dose up to 30 days after last dose (up to week 16)
Population: Safety Analysis Set (SAF) consisted of all participants who took at least 1 dose of IP.
Measure: Number; unit: participants
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 83 | 165
participants | 18 | 58

3. Secondary Outcome: Change From Baseline to Week 12 in Post Void Residual (PVR) Volume
Description: PVR was assessed by ultrasonography.
Time Frame: Baseline, week 12
Population: SAF population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 34 | 144
milliliter | -2.7 (26.3) | -1.3 (24.5)

4. Secondary Outcome: Change From Baseline in Mean Number of Grade 3 or 4 Patient Perception of Intensity of Urgency Scale (PPIUS) Urgency Episodes Per 24 Hours
Description: Urgency was defined as a complaint of a sudden, compelling desire to pass urine, which was difficult to defer. An urgency episode was defined as any micturition or incontinence episode with a severity of grade 3 or 4, assessed by participants based on the PPIUS, where grade 0 = No urgency; grade 1 = Mild urgency; grade 2 = Moderate urgency, could delay voiding a short while; grade 3 = Severe urgency, could not delay voiding; grade 4 = Urge incontinence, leaked before arriving to the toilet. The mean number of urgency episodes (grade 3 and/or 4) per day was calculated as the average number of times a participant recorded an urgency episode (grade 3 and/or 4) with or without incontinence per day during the 3-day micturition diary period.
Time Frame: Baseline and weeks 4, 8, and 12
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: urgency episodes per 24 hours
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 77 | 159
urgency episodes per 24 hours
  Change at Week 4 | -2.09 (2.35) | -2.53 (5.54)
  Change at Week 8: number analyzed (Participants) | 42 | 157
  Change at Week 8 | -2.66 (2.57) | -2.98 (5.78)
  Change at Week 12: number analyzed (Participants) | 36 | 147
  Change at Week 12 | -2.57 (1.92) | -3.55 (5.75)
Statistical Analysis 1: Comparison: Mirabegron 25 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — RMA: CFB as response, TG, visit (week 4, 8 and 12), pooled site, sex and interaction between TG and visit as fixed effects and mean (SD) number of grade 3 or 4 (PPIUS) urgency episodes per 24 hours at baseline as covariate; LS Mean = -2.62, 95% CI 2-sided [-3.25 to -1.99], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Mirabegron 50 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS Mean = -2.47, 95% CI 2-sided [-2.93 to -2.02], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Mirabegron 25 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS Mean = -3.13, 95% CI 2-sided [-3.96 to -2.30], Standard Error of Mean 0.42
Statistical Analysis 4: Comparison: Mirabegron 50 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS Mean = -2.93, 95% CI 2-sided [-3.39 to -2.47], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Mirabegron 25 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS Mean = -3.47, 95% CI 2-sided [-4.37 to -2.56], Standard Error of Mean 0.46
Statistical Analysis 6: Comparison: Mirabegron 50 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 4, analysis 1]; LS Mean = -3.59, 95% CI 2-sided [-4.06 to -3.12], Standard Error of Mean 0.24

5. Secondary Outcome: Change From Baseline in Mean Number of Daytime Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as an episode with any involuntary loss of urine. Daytime was defined as time between waking up in the morning and going to sleep later the same day or next day. The mean number of incontinence episodes was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and at various specified time-intervals.
Time Frame: Baseline and weeks 4, 8, and 12
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: incontinence episodes per 24 hours
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 77 | 159
incontinence episodes per 24 hours
  Change at Week 4 | -0.48 (1.82) | -0.77 (2.47)
  Change at Week 8: number analyzed (Participants) | 42 | 157
  Change at Week 8 | -1.06 (1.85) | -0.89 (2.59)
  Change at Week 12: number analyzed (Participants) | 36 | 147
  Change at Week 12 | -1.03 (1.77) | -0.97 (2.63)
Statistical Analysis 1: Comparison: Mirabegron 25 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — RMA: CFB as response, TG, visit (week 4, 8 and 12), pooled site, sex and the interaction between TG and visit as fixed effects and mean number of daytime incontinence episodes per 24 hours at baseline as covariate; LS Mean = -0.66, 95% CI 2-sided [-0.88 to -0.44], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Mirabegron 50 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; LS Mean = -0.81, 95% CI 2-sided [-0.97 to -0.65], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Mirabegron 25 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; LS Mean = -0.88, 95% CI 2-sided [-1.17 to -0.58], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Mirabegron 50 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; LS Mean = -0.94, 95% CI 2-sided [-1.10 to -0.78], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Mirabegron 25 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; LS Mean = -1.03, 95% CI 2-sided [-1.35 to -0.71], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Mirabegron 50 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; LS Mean = -0.98, 95% CI 2-sided [-1.14 to -0.81], Standard Error of Mean 0.09

6. Secondary Outcome: Change From Baseline in Mean Number of Nighttime Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as an episode with any involuntary loss of urine. Nightime was defined as time between between going to sleep on a day and waking up on the same or next day. The mean number of incontinence episodes was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and at various specified time-intervals.
Time Frame: Baseline and weeks 4, 8, and 12
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: incontinence episodes per 24 hours
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 77 | 159
incontinence episodes per 24 hours
  Change at Week 4 | -0.37 (1.11) | -0.47 (3.06)
  Change at Week 8: number analyzed (Participants) | 42 | 157
  Change at Week 8 | -0.67 (1.50) | -0.45 (3.05)
  Change at Week 12: number analyzed (Participants) | 36 | 147
  Change at Week 12 | -0.42 (0.91) | -0.54 (3.18)
Statistical Analysis 1: Comparison: Mirabegron 25 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — RMA: CFB as response, TG, visit (week 4, 8 and 12), pooled site, sex and the interaction between TG and visit as fixed effects and mean number of nighttime incontinence episodes per 24 hours at baseline as covariate; LS Mean = -0.48, 95% CI 2-sided [-0.58 to -0.37], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Mirabegron 50 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 6, analysis 1]; LS Mean = -0.46, 95% CI 2-sided [-0.53 to -0.38], Standard Error of Mean 0.04
Statistical Analysis 3: Comparison: Mirabegron 25 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 6, analysis 1]; LS Mean = -0.53, 95% CI 2-sided [-0.67 to -0.39], Standard Error of Mean 0.07
Statistical Analysis 4: Comparison: Mirabegron 50 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 6, analysis 1]; LS Mean = -0.45, 95% CI 2-sided [-0.52 to -0.37], Standard Error of Mean 0.04
Statistical Analysis 5: Comparison: Mirabegron 25 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 6, analysis 1]; LS Mean = -0.53, 95% CI 2-sided [-0.68 to -0.38], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Mirabegron 50 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 6, analysis 1]; LS Mean = -0.52, 95% CI 2-sided [-0.60 to -0.45], Standard Error of Mean 0.04

7. Secondary Outcome: Change From Baseline in Mean Number of Urge Incontinence Episodes Per 24 Hours
Description: An incontinence episode was defined as an episode with any involuntary loss of urine. The mean number of urge incontinence episodes per 24 hours was determined using the patient diary data recorded by the participant in the 7 days prior to baseline visit and at various specified time-intervals.
Time Frame: Baseline and weeks 4, 8, and 12
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: urge incontinence episodes per 24 hours
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 77 | 159
urge incontinence episodes per 24 hours
  Change at Week 4 | -0.67 (1.71) | -1.18 (5.02)
  Change at Week 8: number analyzed (Participants) | 42 | 157
  Change at Week 8 | -1.15 (2.38) | -1.25 (5.06)
  Change at Week 12: number analyzed (Participants) | 36 | 147
  Change at Week 12 | -0.92 (1.71) | -1.36 (5.23)
Statistical Analysis 1: Comparison: Mirabegron 25 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — RMA: CFB as response, treatment group, visit (week 4, 8 and 12), pooled site, sex and the interaction between treatment group and visit as fixed effects and mean number of urge incontinence episodes per 24 hours at baseline as covariate; LS Mean = -1.10, 95% CI 2-sided [-1.31 to -0.90], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Mirabegron 50 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean = -1.11, 95% CI 2-sided [-1.25 to -0.96], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Mirabegron 25 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean = -1.26, 95% CI 2-sided [-1.53 to -0.99], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Mirabegron 50 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean = -1.20, 95% CI 2-sided [-1.34 to -1.05], Standard Error of Mean 0.07
Statistical Analysis 5: Comparison: Mirabegron 25 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean = -1.25, 95% CI 2-sided [-1.54 to -0.96], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Mirabegron 50 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 7, analysis 1]; LS Mean = -1.27, 95% CI 2-sided [-1.42 to -1.12], Standard Error of Mean 0.08

8. Secondary Outcome: Change From Baseline in OAB Symptom Score (OABSS)
Description: The OABSS questionnaire was a questionnaire completed by participants with 4 questions regarding their OAB symptoms: Daytime Frequency ("How many times do you typically urinate from waking in the morning until sleeping at night?" where scores range from 0-2), Nighttime Frequency ("How many times do you typically wake up to urinate from sleeping at night until waking in the morning?" where scores range from 0-3), Urgency ("How often do you have a sudden desire to urinate, which is difficult to defer?" where scores range from 0-5), Urgency Incontinence ("How often do you leak urine because you cannot defer the sudden desire to urinate?" where scores range from 0-5). The total score ranges from 0 to 15 with higher score indicating more symptoms.
Time Frame: Baseline and weeks 4, 8, and 12
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 80 | 155
scores on a scale
  Change at Week 4 | -2.91 (2.85) | -3.01 (2.85)
  Change at Week 8: number analyzed (Participants) | 44 | 152
  Change at Week 8 | -5.34 (2.69) | -4.29 (3.01)
  Change at Week 12: number analyzed (Participants) | 37 | 140
  Change at Week 12 | -6.19 (2.72) | -5.43 (3.04)
Statistical Analysis 1: Comparison: Mirabegron 25 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — RMA: CFB as response, TG, visit (week 4, 8 and 12), pooled site, sex and the interaction between TG and visit as fixed effects and mean number of OABSS at baseline as covariate; LS Mean = -2.97, 95% CI 2-sided [-3.50 to -2.43], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Mirabegron 50 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean = -3.05, 95% CI 2-sided [-3.44 to -2.65], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Mirabegron 25 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean = -5.09, 95% CI 2-sided [-5.80 to -4.39], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: Mirabegron 50 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean = -4.30, 95% CI 2-sided [-4.70 to -3.90], Standard Error of Mean 0.20
Statistical Analysis 5: Comparison: Mirabegron 25 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean = -6.01, 95% CI 2-sided [-6.78 to -5.24], Standard Error of Mean 0.39
Statistical Analysis 6: Comparison: Mirabegron 50 mg; Week 12; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean = -5.40, 95% CI 2-sided [-5.82 to -4.98], Standard Error of Mean 0.21

9. Secondary Outcome: Change From Baseline in Mean Number of Micturition Per 24 Hours
Description: as for outcome 1
Time Frame: Baseline and weeks 4 and 8
Population: FAS population with available data at specified time point.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Mirabegron 25 mg | Mirabegron 50 mg
Number analyzed (Participants) | 77 | 159
micturitions per 24 hours
  Change at Week 4 | -2.06 (2.64) | -2.44 (4.62)
  Change at Week 8: number analyzed (Participants) | 42 | 157
  Change at Week 8 | -2.65 (2.55) | -3.01 (4.76)
Statistical Analysis 1: Comparison: Mirabegron 25 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — RMA: CFB as response, TG, visit (week 4, 8), pooled site, sex and the interaction between TG and visit as fixed effects and mean number of micturitions per 24 hours at baseline as covariate; LS Mean = -1.97, 95% CI 2-sided [-2.73 to -1.21], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Mirabegron 50 mg; Week 4; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 9, analysis 1]; LS Mean = -2.36, 95% CI 2-sided [-2.90 to -1.81], Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Mirabegron 25 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 9, analysis 1]; LS Mean = -3.20, 95% CI 2-sided [-4.20 to -2.20], Standard Error of Mean 0.51
Statistical Analysis 4: Comparison: Mirabegron 50 mg; Week 8; Test type: Superiority — Statistical testing was conducted using 2-sided at a significance level of 0.05; p < 0.001, MMRM — [p-value comment as in outcome 9, analysis 1]; LS Mean = -2.92, 95% CI 2-sided [-3.47 to -2.37], Standard Error of Mean 0.28

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after last dose (up to Week 16)
Description: SAF consisted of all participants who took at least 1 dose of IP.
Groups:
- Mirabegron 25 mg (Never Up-titrated): Participants who received single oral dose of mirabegron 25 mg tablet once daily, at the same time after a meal for a duration of 12 weeks and were never up-titrated to receive Mirabegron 50 mg.
- Mirabegron 25 mg (Later Up-titrated to 50 mg): Participants received single oral dose of mirabegron 25 mg tablet once daily, at the same time after a meal until week 4 or 8 and were up-titrated to receive Mirabegron 50 mg until week 12.
- Mirabegron 50 mg (Up-titrated From 25 mg): Participants who were up-titrated from mirabegron 25 mg received single oral dose of Mirabegron 50 mg tablet once daily, at the same time after a meal from week 4 or 8 until week 12.
Arm/Group | Mirabegron 25 mg (Never Up-titrated) | Mirabegron 25 mg (Later Up-titrated to 50 mg) | Mirabegron 50 mg (Up-titrated From 25 mg) | Mirabegron 50 mg
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/39 | 0/39 | 0/165
Serious Adverse Events (participants affected / at risk) | 3/44 | 1/39 | 2/39 | 8/165
Other Adverse Events (participants affected / at risk) | 1/44 | 0/39 | 3/39 | 6/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron 25 mg (Never Up-titrated) (N=44) | Mirabegron 25 mg (Later Up-titrated to 50 mg) (N=39) | Mirabegron 50 mg (Up-titrated From 25 mg) (N=39) | Mirabegron 50 mg (N=165)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirabegron 25 mg (Never Up-titrated) (N=44) | Mirabegron 25 mg (Later Up-titrated to 50 mg) (N=39) | Mirabegron 50 mg (Up-titrated From 25 mg) (N=39) | Mirabegron 50 mg (N=165)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT04562090/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT04562090/SAP_001.pdf